CLINICAL TRIAL: NCT06512974
Title: A Feasibility and Efficacy Study of NeuroTrainer Cognitive Training in Students With and Without Attention-Related Difficulties
Brief Title: NeuroTrainer Cognitive Training For Academic Focus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NeuroTrainer (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of California, Davis (Other)
Responsible Party: Principal Investigator, Jeff Nyquist, Chief Science Officer, NeuroTrainer
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R43MH135599-01A1 (NIH)
Record Dates: First submitted 2024-07-10; First posted 2024-07-22 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: ADHD - Combined Type; ADHD Predominantly Inattentive Type; ADHD, Predominantly Hyperactive - Impulsive
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: This study will evaluate the efficacy of NeuroTrainer cognitive training for improving attention and executive function in students with ADHD and sub threshold ADHD, divided into intervention and control groups. Participants, aged 11-17, will be randomly assigned to use NeuroTrainer or receive standard educational activity. Primary outcomes include attention and executive function improvements, while secondary outcomes assess ADHD symptoms and academic performance. Data will be collected at baseline, midpoint, post-intervention and 6-month follow-up.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NeuroTrainer Intervention (Experimental): The NeuroTrainer intervention involves using a VR-based cognitive training program designed to improve attention and executive function in students with ADHD. Participants will engage in 30-minute sessions, approximately three times a week for 12 weeks, performing game-like tasks that integrate physical activity and adapt to their performance level.
  Interventions: Behavioral: NeuroTrainer
- Control Condition (No Intervention): The control condition involves students receiving standard educational interventions without the use of NeuroTrainer. These activities include regular classroom instruction and typical academic tasks designed to support learning, without the additional cognitive training provided by the VR program.

INTERVENTIONS:
Behavioral: NeuroTrainer — Virtual reality based cognitive training
  Arms: NeuroTrainer Intervention

SUMMARY:
This clinical trial aims to evaluate the feasibility and efficacy of NeuroTrainer cognitive training in improving attentional and executive control functions in students with and without attention-related difficulties.

DETAILED DESCRIPTION:
The goal of this clinical trial is to test the feasibility and efficacy of NeuroTrainer cognitive training in improving attentional and executive control function in students with and without attention-related difficulties. The main questions it aims to answer are (1) does NeuroTrainer improve attentional and executive control function, (2) does NeuroTrainer engage the target of ADHD inattention symptoms by identifying the target and demonstrating proximal changes in it, and (3) does NeuroTrainer demonstrate transfer of skill with improvement in academic behaviors. Researchers will compare students who use NeuroTrainer to a control condition to see if the NeuroTrainer intervention produces significant improvements.

Participants in the intervention group will engage in virtual reality (VR) sessions which include physical activity and cognitive training. Cognitive training will maximize time at performance thresholds and optimize for variability in task dynamics and demands.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic criteria met ADHD for any ADHD presentation type, with severity ratings of subthreshold, moderate or severe
* Estimated IQ of 80 or greater
* Between 11-17 years of age

Exclusion Criteria:

* Presence of suicidality
* Presence of psychotic disorders
* Visual or hearing impairment
* Presence of severe depression

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 155 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
NIH Toolbox Flanker Inhibitory Control and Attention Test (RT) | Week 1, Month 2, Month 3, Month 9
  This test is designed to evaluate an individual's ability to concentrate their attention while inhibiting automatic response tendencies that could potentially hinder goal achievement. The assessment has demonstrated changes in ADHD cases (Buzy, et al., 2009) and may be sensitive to treatment effects (Epstein et al., 2011). The test will take approximately 3 minutes to complete. This is the reaction time (RT) outcome from this assessment.
NIH Toolbox Flanker Inhibitory Control and Attention Test (IIV-RT) | Week 1, Month 2, Month 3, Month 9
  This test is designed to evaluate an individual's ability to concentrate their attention while inhibiting automatic response tendencies that could potentially hinder goal achievement. The assessment has demonstrated changes in ADHD cases (Buzy, et al., 2009) and may be sensitive to treatment effects (Epstein et al., 2011). The test will take approximately 3 minutes to complete. This is the intraindividual variability of RT (IIV-RT) outcome from this assessment.
NIH Toolbox Flanker Inhibitory Control and Attention Test (% Correct) | Week 1, Month 2, Month 3, Month 9
  This test is designed to evaluate an individual's ability to concentrate their attention while inhibiting automatic response tendencies that could potentially hinder goal achievement. The assessment has demonstrated changes in ADHD cases (Buzy, et al., 2009) and may be sensitive to treatment effects (Epstein et al., 2011). The test will take approximately 3 minutes to complete. This is the percent correct outcome from this assessment.
NIH Toolbox Dimensional Change Card Sort Test (% Correct) | Week 1, Month 2, Month 3, Month 9
  This test aims to measure an individual's capacity to switch between multiple aspects of a strategy or task. The test takes approximately 4 minutes to complete. This is the percent correct outcome from this assessment.
NIH Toolbox Dimensional Change Card Sort Test (Omissions) | Week 1, Month 2, Month 3, Month 9
  This test aims to measure an individual's capacity to switch between multiple aspects of a strategy or task. The test takes approximately 4 minutes to complete. This is the omissions outcome from this assessment.
NIH Toolbox Dimensional Change Card Sort Test (RT) | Week 1, Month 2, Month 3, Month 9
  This test aims to measure an individual's capacity to switch between multiple aspects of a strategy or task. The test takes approximately 4 minutes to complete. This is the response time (RT) outcome from this assessment.
NIH Toolbox Dimensional Change Card Sort Test (IIV-RT) | Week 1, Month 2, Month 3, Month 9
  This test aims to measure an individual's capacity to switch between multiple aspects of a strategy or task. The test takes approximately 4 minutes to complete. This is the intraindividual variability of RT (IIV-RT) outcome from this assessment.
NIH Toolbox List Sorting Working Memory Test | Week 1, Month 2, Month 3, Month 9
  This test serves as an evaluation of an individual's working memory capabilities. Participants will be presented with different stimuli visually and audibly, and they will be asked to recall and sequence them accordingly. The test takes approximately 7 minutes to complete.
NIH Toolbox Pattern Comparison Processing Speed Test | Week 1, Month 2, Month 3, Month 9
  This is an assessment of processing speed. Participants are asked to quickly determine whether two stimuli are the same or not the same. The test takes approximately 4 minutes to complete.

SECONDARY OUTCOMES:
ADHD Rating Scale-5 (ADHD:RS-5) - Inattention Subscale | Week 1, Month 2, Month 3, Month 9
  The investigators will assess the symptoms of ADHD by utilizing the parent and teacher ADHD Rating Scale-5 (ADHD:RS-5) Inattention Subscale, using two academic teachers and one parent for each participant. This 9-item subscale is specifically designed to evaluate the core ADHD symptoms of Inattention. By incorporating the perspectives of both teachers and parents, the investigators aim to obtain a comprehensive understanding of the participants' ADHD symptoms across settings. ADHD:RS-5: will be completed by prior school year teachers if the student has been in the class for less than 2 months. Higher scores represent a higher frequency of symptoms and this a worse outcome. For each item, "0" is the minimum and "3" is the maximum value.
ADHD Rating Scale-5 (ADHD:RS-5) - Impulsivity/Hyperactivity Subscale | Week 1, Month 2, Month 3, Month 9
  The investigators will assess the symptoms of ADHD by utilizing the parent and teacher ADHD Rating Scale-5 (ADHD:RS-5) Impulsivity/Hyperactivity Subscale, using two academic teachers and one parent for each participant. This 9-item subscale is specifically designed to evaluate the core ADHD symptoms of Impulsivity/Hyperactivity. By incorporating the perspectives of both teachers and parents, the investigators aim to obtain a comprehensive understanding of the participants' ADHD symptoms across settings. ADHD:RS-5: will be completed by prior school year teachers if the student has been in the class for less than 2 months. Higher scores represent a higher frequency of symptoms and this a worse outcome. For each item, "0" is the minimum and "3" is the maximum value.
Academic Performance Rating Scale (APRS) | Week 1, Month 2, Month 3, Month 9
  The 19-item Academic Performance Rating Scale (APRS; DuPaul et al.,1991) evaluates student academic performance and is ecologically valid due to (1) assessing in real classroom environments, mirroring academic challenges and behaviors, (2) evaluated by teachers who gain insights into students' academic performance beyond standard tests, and (3) encompassing aspects of academic abilities including behavior, productivity, and work accuracy. This scale has a high test-retest reliability (2-week test-retest=.93-.95; α=.94-.95). Higher scores indicate better academic functioning and impulse control in school. For each item, "1" is the minimum and "5" is the maximum value.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Nyquist, Ph.D., Principal Investigator — NeuroTrainer
Locations (3):
- United States (3):
  - Marquette Senior High School, Marquette, Michigan
  - Westside High School, Omaha, Nebraska
  - One City Schools, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No